CLINICAL TRIAL: NCT00558142
Title: Mechanisms for the Effect of Acetylcysteine on Renal Function After Exposure to Radiographic Contrast Material
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: NAC0606; NRES reference: 07/MRE00/64; EudraCT reference: 2006; 003509-18
Record Dates: First submitted 2007-11-13; First posted 2007-11-14 (Estimated); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2021-04

CONDITIONS: Radiocontrast-induced Nephropathy
Keywords: contrast nephropathy; radiocontrast-induced nephropathy; chronic kidney disease; acetylcysteine; clinical study
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Acetylcysteine; N-monoacetylcystine; iodixanol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Active Comparator): Healthy volunteers will be randomised to receive either placebo capsules PO plus an infusion of normal saline, acetylcysteine capsules PO plus an infusion of normal saline or placebo capsules PO plus an IV infusion of acetylcysteine in normal saline
  Interventions: Drug: Acetylcysteine
- 2 (Active Comparator): Volunteers with CKD III will be randomised to receive either placebo capsules PO plus an infusion of normal saline, acetylcysteine capsules PO plus an infusion of normal saline or placebo capsules PO plus an IV infusion of acetylcysteine in normal saline
  Interventions: Drug: Acetylcysteine
- 3 (Active Comparator): Healthy volunteers will receive a single IV dose of 100mls Visipaque 320 (iodixanol, equivalent to 320 mg iodine/ml). They will then be randomised to receive either placebo capsules PO plus an infusion of normal saline, acetylcysteine capsules PO plus an infusion of normal saline or placebo capsules PO plus an IV infusion of acetylcysteine in normal saline
  Interventions: Drug: Acetylcysteine; Drug: Visipaque 320
- 4 (Active Comparator): Volunteers with CKD III will receive Visipaque 320 during coronary angiography. They will have been randomised to receive either placebo capsules PO plus an infusion of normal saline, acetylcysteine capsules PO plus an infusion of normal saline or placebo capsules PO plus an IV infusion of acetylcysteine in normal saline
  Interventions: Drug: Acetylcysteine; Drug: Visipaque 320

INTERVENTIONS:
Drug: Acetylcysteine — Participants will receive packs of either 8 placebo capsules or 8 acetylcysteine (600mg) capsules. They will be asked to take 2 tablets at 08.00 and 22.00 on the day before the study and the day of the study. On the day of the study participants will receive an IV infusion of either normal saline or acetylcysteine (200mg/kg)
  Other Names: Parvolex
Drug: Visipaque 320 — 100mls IV dose as single dose
  Other Names: Iodixanol
  Arms: 3
Drug: Visipaque 320 — The dose of Visipaque will be administered by the consultant cardiologist performing the coronary angiography
  Other Names: Iodixanol
  Arms: 4

SUMMARY:
Millions of people receive radiographic contrast material for investigations like CT and coronary angiography. While considered safe in healthy patients, it can cause acute renal impairment. This is termed radiocontrast-induced nephropathy (RCIN) and is generally defined as an increase in serum creatinine over baseline of more than 25% or 0.5 mg/dL (44.2 μmol/l) within 48 hrs. RCIN occurs in less than 2% of patients with normal renal function but is more common in patients with pre-existing renal damage.

The pathophysiology of RCIN is unclear. Possible mechanisms involve 1) reduced renal blood flow leading to acute tubular necrosis and 2) direct renal tubular injury by oxygen free radicals. Current prevention strategies focus on increasing renal blood flow and reducing oxidative stress. Patients at risk of RCIN currently receive fluids, a low dose of contrast, and variable and unproven doses of acetylcysteine.

The evidence for acetylcysteine administration is unclear. A RCIN consensus working group reported in the American Journal of Cardiology in September 2006 that "N-acetylcysteine is not consistently effective in reducing the risk for contrast-induced nephropathy". The perception of a benefit from acetylcysteine administration that is unproven has disadvantages as some clinicians report giving larger amounts of radio-contrast to patients who have received acetylcysteine since they believe that it prevents RCIN. There is a need to determine how acetylcysteine might prevent RCIN and to identify the appropriate dose and route of administration.

Since acetylcysteine is a vasodilator as well as an antioxidant, it may work in two distinct ways, by preventing reduction in renal blood flow (RBF) or contrast-induced oxidative damage. Previous studies have used changes in serum creatinine. In addition to being an insensitive marker of altered renal function, if contrast causes renal vasoconstriction and acetylcysteine vasodilatation, changes in serum creatinine will not be the ideal marker of effect. Finally the optimum dose and route of acetylcysteine administration is unclear, as illustrated by studies using a variety of doses and routes.

We propose to study the mechanism of effects of acetylcysteine on healthy and diseased kidneys, both unstressed and stressed by radiocontrast administration. We hypothesise that acetylcysteine may exert a renoprotective effect in RCIN by a renal vasodilatation and/or antioxidant mechanism.

DETAILED DESCRIPTION:
In this study we will test the hypothesis that acetylcysteine exerts a renoprotective effect in RCIN by an antioxidant and/or renal vasodilator mechanism.

We will take a structured 4-part approach, using randomised controlled cross-over studies to assess the effect of acetylcysteine on renal function in both normal and diseased kidneys, and then the effect of contrast on normal kidneys, with and without acetylcysteine treatment. We will also perform a parallel-group randomised controlled trial of angiography on CKD patients with and without acetylcysteine treatment. The four groups will be studied simultaneously. As per the decision of the MHRA, this study is a phase IV trial of an authorized medication rather than a phase I trial.

The study will be performed simultaneously in four groups of participants, studying:

1. healthy volunteers receiving acetylcysteine PO, acetylcysteine IV, or placebo
2. volunteers with stage III CKD receiving acetylcysteine PO, acetylcysteine IV, or placebo
3. healthy volunteers receiving radiographic contrast plus acetylcysteine PO, acetylcysteine IV, or placebo
4. patients with stage III CKD receiving radiographic contrast for elective coronary angiography plus acetylcysteine PO, acetylcysteine IV, or placebo.

The study will be performed in the Wellcome Trust Clinical Research Facility at the Royal Infirmary of Edinburgh (RIE). Volunteers will be paid £120 to cover travelling and other expenses for each study arm.

STUDIES 1 AND 2 These studies will assess the effect of acetylcysteine alone in healthy volunteers or in volunteers with stage III CKD. Volunteers will be randomised to a three-way, cross-over, double-blind comparison of matched placebo with oral and intravenous regimens of acetylcysteine. The primary outcome will be change in RBF (measured as para-aminohippuric acid [PAH] clearance). In addition, GFR (measured as inulin clearance), tubular function (fractional excretion of potassium and sodium), oxidative balance (total oxidative capacity, plasma and urinary isoprostanes), and plasma and urinary endothelin-1 will be assayed. The pharmacokinetics of acetylcysteine will be measured to compare IV and PO regimens.

Volunteers will be randomised to receive on three occasions, separated by at least two weeks, one of:

A) placebo capsules PO, plus an IV infusion acetylcysteine in normal saline. B) acetylcysteine capsules PO, plus an infusion of normal saline. C) placebo capsules PO, plus an infusion of normal saline.

DOSE JUSTIFICATION There are currently no data to guide choice of an optimum oral or IV acetylcysteine regimen. This study will assess the effects of an IV and an oral dose of acetylcysteine (IV 200mg/kg; PO 68.6 mg/kg) that are very similar to those currently used in clinical practice. The oral dose is expected to produce a plasma concentration much lower than the IV dose; however, it is believed that a first pass effect after oral administration may increase conversion in the liver of acetylcysteine into cysteine and then glutathione, increasing the efficacy of an oral dose. The first clinical trials in RCIN used an arbitrary low dose oral regimen of acetylcysteine - 600mg twice a day (BD) for 2 days, starting the day before dye administration (total dose 2.4 g, 34.3 mg/kg in a 70kg patient). Recent studies have used higher total doses of up to 1500mg BD for 2 days (total dose 6 g, 85.7 mg/kg in a 70kg patient). IV regimens have also been assessed since they have been proposed to be effective when started on the same day as the dye administration, rather than the day before. The first trial used a dose similar to that used for early treatment of paracetamol-induced hepatotoxicity - 150 mg/kg over 30 min, then 50mg/kg over 4 hrs (total dose 200 mg/kg) - and reported less nephropathy. Other studies used lower doses (eg. 500 mg over 15 mins [7.1 mg/kg in 70 kg patient] or 1000 mg twice, before and after the procedure, [28.5 mg/kg in 70kg patient]) and did not find any benefit. Overall, the choice of acetylcysteine regimen for previous studies seems to have been based on ease and prior practice in paracetamol poisoning rather than knowledge of acetylcysteine's effects on the kidney.

We have chosen a revised IV high dose regimen derived from PK data published by Dr L Prescott after Monte Carlo simulations (Dr R Thanacoody, Consultant Clinical Pharmacologist, Edinburgh Royal infirmary, unpublished) for 2 reasons:

1. the RCT that showed benefit with IV acetylcysteine used a high dose regimen similar to that used for paracetamol poisoning (150 mg/kg over 30 min, then 50 mg/kg over 4 hrs). The subsequent negative studies used much lower doses, suggesting that IV acetylcysteine may need to be given in high doses.
2. the high peak plasma concentration that results from the rapid initial infusion of acetylcysteine for paracetamol poisoning produces nausea in about 40% of patients and anaphylactoid reactions in about 20%. Although these reactions are routine and normally easily treated, it is important to reduce the rate of such reactions in study participants. The revised regimen provides a similar amount of acetylcysteine but administers it more evenly across 7 hours, producing a lower peak acetylcysteine concentration and a lower likelihood of nausea and anaphylactoid reactions (Dr R Thanacoody, unpublished).

The choice of oral acetylcysteine regimen is necessarily arbitrary. We will use 1200 mg since there is some evidence that it is more effective than the more usually administered 600 mg.

STUDY 3 This study will assess the effect of acetylcysteine on renal function in healthy volunteers receiving a single IV 100ml dose of Visipaque 320 (iodixanol, equivalent to 320 mg iodine/ml), an iso-osmolar non-ionic radio-contrast agent, via a peripheral cannula. We chose this dose because 100 mls are routinely used in the Royal Infirmary for coronary angiography in CKD patients (Radiology Dept, personal communication). Larger doses of up to 400 ml are then used if an angioplasty is subsequently required. Such doses fall within the doses recommended in the summary of product characteristics, Martindale, and the literature. The safety profile of such doses in healthy adults is excellent; in patients with CKD, iodixanol is at least as safe as other contrast agents.

Volunteers will be randomised in this study to a three-way, cross-over, double-blind comparison of placebo with oral and intravenous regimens of acetylcysteine. They will not receive coronary angiography, just the intravenous contrast.

We will study healthy volunteers in order to identify the effects of NAC and contrast on healthy kidneys. This will provide baseline data for interpreting the studies in CKD patients. In addition, while healthy patients rarely get RCIN after contrast administration, the currently used marker of RCIN (raised serum creatinine) is a crude measure of renal dysfunction - since GFR will only fall after renal RBF has been substantially reduced for a significant period of time. It is likely that small sub-clinical changes will occur in healthy patients that will help determine how contrast and NAC affect the kidney.

STUDY 4 This study will assess the effect of acetylcysteine on renal function in stable stage III CKD patients receiving 100 ml of iodixanol during routine coronary angiography. Recruited patients will not receive multiple angiographies so study 4 will not be a crossover comparison but a randomised controlled study of oral acetylcysteine vs. IV acetylcysteine vs. placebo. Results from studies 1-3 will inform the analysis and interpretation of this study.

MEASUREMENTS OF RENAL FUNCTION Most previous RCTs have measured changes in serum creatinine concentration rather than any direct measures of renal failure. Serum creatinine concentration can provide information on GFR. However, it is not accurate since it is affected by diet, aging and muscle mass. Furthermore, acetylcysteine also lowers serum creatinine concentration itself, suggesting that the lower creatinine noted in the RCTs may not actually reflect improved renal function. GFR is the best marker of global renal function. It can be directly measured using the 51Cr-EDTA method but this is a complicated technique. We will use an alternative method by measuring plasma clearance of inulin. Serum cystatin C concentration may be a better marker of GFR than creatinine. Cystatin C is a small cysteine protease that is secreted at a fixed rate by all nucleated cells and is not affected by diet or muscle mass. In RCIN, serum cystatin concentration peaks and normalises more rapidly than creatinine. We will measure cystatin C in these patients to assess whether it would be a better marker of GFR in future RCTs.

Changes in renal blood flow after acetylcysteine and/or contrast administration will be assessed by measuring plasma PAH clearance. Endothelin-1 (ET-1) is a potent endogenous vasoconstrictor and increased urinary ET-1 has been associated with the development of RCIN. Changes in renal ET-1 production will be measured following acetylcysteine and/or contrast by measuring ET-1 concentrations in plasma and urine and calculating its fractional excretion. Renal tubular function will be assessed by measuring the kidney's fractional excretion of sodium and potassium. Reductions in fractional excretion of these ions will supply information on renal perfusion and tubular function, and have been noted previously in RCIN. We will also measure urine levels of proteins released from damaged tubular cells.

Since acetylcysteine should alter oxidative state, we will measure the oxidative balance through assays for plasma and urinary isoprostanes, plasma N-acetylcysteine, peripheral blood cell glutathione, and total antioxidant capacity.

ADMINISTRATION OF ORAL ACETYLCYSTEINE/PLACEBO Participants will receive 3 blister packs of acetylcysteine or placebo capsules and be asked to take the appropriate capsules at 08.00 and 20.00 on the day before the study day (Day 1; Day 2 being the day spent in the CRF). They will also be asked to drink an extra 500ml of water to ensure adequate hydration. Hard capsules containing acetylcysteine 600 mg or matched placebo (Lactose PhEur 600 mg) will be prepared by Tayside Pharmaceuticals, Dundee, and packaged in patient packs of 8 capsules. The capsules will be delivered to the hospital pharmacy and supplied to participants according to the randomized allocation order.

INTRAVENOUS ADMINISTRATION OF DRUGS Inulin and PAH will be administered through a 20G venous cannula inserted into the forearm. Inulin and PAH will be infused at a constant infusion rate throughout the 8 hour study period. Acetylcysteine/placebo will be administered through a second 20G venous cannula inserted into the same forearm. We will use the intravenous acetylcysteine preparation currently used in the Royal Infirmary of Edinburgh (Parvolex, UCB Pharma Limited). Placebo will be sodium chloride solution for infusion. Active or placebo infusions will be prepared by the Clinical Research Facility on each study day according to the randomized allocation order.

VENOUS BLOOD SAMPLING Blood samples will be obtained via a 17G venous cannula inserted into the other forearm. Samples will be taken hourly on 10 occasions from -1h (beginning of the inulin/PAH infusion) to 8h; a total of 120 mls will be taken. Blood will also be sampled at 24h (09.00 on day 3) and 72h 09.00 on day 5); 24 ml at each time.

URINE SAMPLING 40ml urine samples will be taken after voiding every two hours, from 0h to 8h on day 1, and again at 24h (09.00 on day 3) and 72h (09.00 on day 5). Participants will be asked to void urine on waking on days 3 and 5. At the end of each study, the venous cannulae will be removed and haemostasis confirmed. Subjects will be provided with toast and a warm beverage and observed for 30 minutes before leaving the unit.

ELIGIBILITY:
Inclusion Criteria:

* Study 1 and 3: Healthy male volunteers over 45 years of age with BMI between 22 and 40.
* Study 2: Male volunteers with CKD III with BMI between 22 and 40.
* Study 4: Male patients over 45 year of age with stable CKD III and BMI between 22 and 40, undergoing elective coronary angiography.

Exclusion Criteria for studies 1 and 3:

* Lack of informed consent
* Age <46 years
* Current involvement in a clinical trial
* Clinically significant co-morbidity: heart failure, hypertension, known hyperlipidaemia, diabetes mellitus, coagulopathy, peripheral vascular disease, or bleeding disorder
* thyroid disease, myasthenia gravis, asthma, atopy, or a history of allergy/sensitivity to acetylcysteine or contrast medium
* current intake of prescription medicines, in particular beta blockers
* recent infective/inflammatory condition
* blood donation during the preceding three months

Exclusion criteria for studies 2 and 4:

* Lack of informed consent
* Age <46 years
* Current involvement in a clinical trial
* Thyroid disease, myasthenia gravis, asthma, atopy, or a history of allergy/sensitivity to acetylcysteine or contrast medium
* Recent infective/inflammatory condition
* Blood donation during the preceding three months

Min Age: 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2008-02; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Eddleston, MA PhD MCRP, Principal Investigator — University of Edinburgh
Locations (1):
- Clinical Research Facility, Royal Infirmary Edinburgh, Edinburgh, Midlothian, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Parfrey P. The clinical epidemiology of contrast-induced nephropathy. Cardiovasc Intervent Radiol. 2005;28 Suppl 2:S3-11. doi: 10.1007/s00270-005-0196-8. PMID 16419277
- [Background] Gleeson TG, Bulugahapitiya S. Contrast-induced nephropathy. AJR Am J Roentgenol. 2004 Dec;183(6):1673-89. doi: 10.2214/ajr.183.6.01831673. No abstract available. PMID 15547209
- [Background] Stacul F. Reducing the risks for contrast-induced nephropathy. Cardiovasc Intervent Radiol. 2005;28 Suppl 2:S12-8. doi: 10.1007/s00270-005-0197-7. PMID 16419278
- [Background] Marenzi G, Assanelli E, Marana I, Lauri G, Campodonico J, Grazi M, De Metrio M, Galli S, Fabbiocchi F, Montorsi P, Veglia F, Bartorelli AL. N-acetylcysteine and contrast-induced nephropathy in primary angioplasty. N Engl J Med. 2006 Jun 29;354(26):2773-82. doi: 10.1056/NEJMoa054209. PMID 16807414
- [Background] Eddleston M, Goddard J, Bateman N. N-acetylcysteine for contrast nephropathy: more clinical science is required. Arch Intern Med. 2006 Aug 14-28;166(15):1668-9; author reply 1669. doi: 10.1001/archinte.166.15.1668-b. No abstract available. PMID 16908804
- [Derived] Sandilands EA, Cameron S, Paterson F, Donaldson S, Briody L, Crowe J, Donnelly J, Thompson A, Johnston NR, Mackenzie I, Uren N, Goddard J, Webb DJ, Megson IL, Bateman N, Eddleston M. Mechanisms for an effect of acetylcysteine on renal function after exposure to radio-graphic contrast material: study protocol. BMC Clin Pharmacol. 2012 Feb 3;12:3. doi: 10.1186/1472-6904-12-3. PMID 22305183

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Volunteers, no Contrast: Healthy volunteers will be randomised to receive either placebo capsules PO plus an infusion of normal saline, acetylcysteine capsules PO plus an infusion of normal saline or placebo capsules PO plus an IV infusion of acetylcysteine in normal saline
  Acetylcysteine: Participants will receive packs of either 8 placebo capsules or 8 acetylcysteine (600mg) capsules. They will be asked to take 2 tablets at 08.00 and 22.00 on the day before the study and the day of the study. On the day of the study participants will receive an IV infusion of either normal saline or acetylcysteine (200mg/kg)
- CKDIII Patients, no Contrast: Volunteers with CKD III will be randomised to receive either placebo capsules PO plus an infusion of normal saline, acetylcysteine capsules PO plus an infusion of normal saline or placebo capsules PO plus an IV infusion of acetylcysteine in normal saline
  Acetylcysteine: Participants will receive packs of either 8 placebo capsules or 8 acetylcysteine (600mg) capsules. They will be asked to take 2 tablets at 08.00 and 22.00 on the day before the study and the day of the study. On the day of the study participants will receive an IV infusion of either normal saline or acetylcysteine (200mg/kg)
- Healthy Volunteers, With Contrast: Healthy volunteers will receive a single IV dose of 100mls Visipaque 320 (iodixanol, equivalent to 320 mg iodine/ml). They will then be randomised to receive either placebo capsules PO plus an infusion of normal saline, acetylcysteine capsules PO plus an infusion of normal saline or placebo capsules PO plus an IV infusion of acetylcysteine in normal saline
  Acetylcysteine: Participants will receive packs of either 8 placebo capsules or 8 acetylcysteine (600mg) capsules. They will be asked to take 2 tablets at 08.00 and 22.00 on the day before the study and the day of the study. On the day of the study participants will receive an IV infusion of either normal saline or acetylcysteine (200mg/kg)
  Visipaque 320: 100mls IV dose as single dose
- CKD III Patients, With Contrast: Volunteers with CKD III will receive Visipaque 320 during coronary angiography. They will have been randomised to receive either placebo capsules PO plus an infusion of normal saline, acetylcysteine capsules PO plus an infusion of normal saline or placebo capsules PO plus an IV infusion of acetylcysteine in normal saline
  Acetylcysteine: Participants will receive packs of either 8 placebo capsules or 8 acetylcysteine (600mg) capsules. They will be asked to take 2 tablets at 08.00 and 22.00 on the day before the study and the day of the study. On the day of the study participants will receive an IV infusion of either normal saline or acetylcysteine (200mg/kg)
  Visipaque 320: The dose of Visipaque will be administered by the consultant cardiologist performing the coronary angiography
Period: Overall Study
Arm/Group | Healthy Volunteers, no Contrast | CKDIII Patients, no Contrast | Healthy Volunteers, With Contrast | CKD III Patients, With Contrast
Started | 10 | 13 | 8 | 76
Completed | 8 | 8 | 8 | 66
Not Completed | 2 | 5 | 0 | 10

BASELINE CHARACTERISTICS:
Groups:
- CKD III Patients, no Contrast: Volunteers with CKD III will be randomised to receive either placebo capsules PO plus an infusion of normal saline, acetylcysteine capsules PO plus an infusion of normal saline or placebo capsules PO plus an IV infusion of acetylcysteine in normal saline
  Acetylcysteine: Participants will receive packs of either 8 placebo capsules or 8 acetylcysteine (600mg) capsules. They will be asked to take 2 tablets at 08.00 and 22.00 on the day before the study and the day of the study. On the day of the study participants will receive an IV infusion of either normal saline or acetylcysteine (200mg/kg)
- Total: Total of all reporting groups
Arm/Group | Healthy Volunteers, no Contrast | CKD III Patients, no Contrast | Healthy Volunteers, With Contrast | CKD III Patients, With Contrast | Total
Number analyzed (Participants) | 8 | 8 | 8 | 66 | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 3 | 7 | 16
  >=65 years | 5 | 5 | 5 | 59 | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (2) | 57 (3) | 57 (3) | 73 (6) | 69 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 8 | 8 | 8 | 66 | 90
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 8 | 8 | 8 | 65 | 89
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 8 | 8 | 8 | 66 | 90

OUTCOME MEASURES:

1. Primary Outcome: Changes in Renal Blood Flow
Description: Measurement of change in renal blood flow through para-aminohippuric acid (PAH) elimination
Time Frame: 0, 2, 2.25, 2.5, 4, 6, and 8 hrs
Measure: Mean (95% Confidence Interval); unit: h.mL/min
Groups:
- Volunteers With CKD III, no Contrast: Volunteers with CKD III will be randomised to receive either placebo capsules PO plus an infusion of normal saline, acetylcysteine capsules PO plus an infusion of normal saline or placebo capsules PO plus an IV infusion of acetylcysteine in normal saline
  Acetylcysteine: Participants will receive packs of either 8 placebo capsules or 8 acetylcysteine (600mg) capsules. They will be asked to take 2 tablets at 08.00 and 22.00 on the day before the study and the day of the study. On the day of the study participants will receive an IV infusion of either normal saline or acetylcysteine (200mg/kg)
- Healthy Volunteers With Contrast: Healthy volunteers will receive a single IV dose of 100mls Visipaque 320 (iodixanol, equivalent to 320 mg iodine/ml). They will then be randomised to receive either placebo capsules PO plus an infusion of normal saline, acetylcysteine capsules PO plus an infusion of normal saline or placebo capsules PO plus an IV infusion of acetylcysteine in normal saline
  Acetylcysteine: Participants will receive packs of either 8 placebo capsules or 8 acetylcysteine (600mg) capsules. They will be asked to take 2 tablets at 08.00 and 22.00 on the day before the study and the day of the study. On the day of the study participants will receive an IV infusion of either normal saline or acetylcysteine (200mg/kg)
  Visipaque 320: 100mls IV dose as single dose
- Volunteers With CKD III, With Contrast: Patients with CKD III will receive Visipaque 320 during coronary angiography. They will have been randomised to receive either placebo capsules PO plus an infusion of normal saline, acetylcysteine capsules PO plus an infusion of normal saline or placebo capsules PO plus an IV infusion of acetylcysteine in normal saline
  Acetylcysteine: Participants will receive packs of either 8 placebo capsules or 8 acetylcysteine (600mg) capsules. They will be asked to take 2 tablets at 08.00 and 22.00 on the day before the study and the day of the study. On the day of the study participants will receive an IV infusion of either normal saline or acetylcysteine (200mg/kg)
  Visipaque 320: The dose of Visipaque will be administered by the consultant cardiologist performing the coronary angiography
Arm/Group | Healthy Volunteers, no Contrast | Volunteers With CKD III, no Contrast | Healthy Volunteers With Contrast | Volunteers With CKD III, With Contrast
Number analyzed (Participants) | 8 | 8 | 8 | 66
h.mL/min
  IV NAC | 9590.8 [9168.4 to 10013.2] | 5105.4 [4714.0 to 5496.9] | 8529.4 [8096.7 to 8962.1] | 5228.4 [4935.4 to 5521.3]
  PO NAC | 9088.6 [8668.6 to 9508.6] | 4909.3 [4517.8 to 5300.7] | 7648.2 [7213.3 to 8083.2] | 5038.9 [4740.0 to 5337.9]
  No NAC, placebo | 8876.5 [8452.5 to 9300.5] | 4817.3 [4426.0 to 5208.5] | 7612.8 [7185.1 to 8040.6] | 5077.8 [4785.8 to 5369.8]

2. Secondary Outcome: Changes in Glomerular Filtration Rate
Description: Measurement of change in AUC for glomerular filtration rate through inulin elimination
Time Frame: 0, 2, 2.25, 2.5, 4, 6, and 8 hrs
Population: Difference between AUCs for IV NAC and placebo
Measure: Mean (95% Confidence Interval); unit: h*mL/ min/1.73 m²
Arm/Group | Healthy Volunteers, no Contrast | Volunteers With CKD III, no Contrast | Healthy Volunteers With Contrast | Volunteers With CKD III, With Contrast
Number analyzed (Participants) | 8 | 8 | 8 | 65
h*mL/ min/1.73 m² | 29.3 [-27.8 to 86.4] | 5.9 [-30.8 to 42.6] | 146.8 [77.1 to 216.5] | 28.7 [-7.9 to 65.3]

ADVERSE EVENTS:
Description: Adverse events are collected per study (4 reported here - 3 cross-over, 1 parallel group study). Adverse events are reported as per study
Groups:
- Patients With CKD III, With Contrast: Patients with CKD III will receive Visipaque 320 during coronary angiography. They will have been randomised to receive either placebo capsules PO plus an infusion of normal saline, acetylcysteine capsules PO plus an infusion of normal saline or placebo capsules PO plus an IV infusion of acetylcysteine in normal saline
  Acetylcysteine: Participants will receive packs of either 8 placebo capsules or 8 acetylcysteine (600mg) capsules. They will be asked to take 2 tablets at 08.00 and 22.00 on the day before the study and the day of the study. On the day of the study participants will receive an IV infusion of either normal saline or acetylcysteine (200mg/kg)
  Visipaque 320: The dose of Visipaque will be administered by the consultant cardiologist performing the coronary angiography
Arm/Group | Healthy Volunteers, no Contrast | Volunteers With CKD III, no Contrast | Healthy Volunteers, With Contrast | Patients With CKD III, With Contrast
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/66
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 6/66
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 15/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Volunteers, no Contrast (N=8) | Volunteers With CKD III, no Contrast (N=8) | Healthy Volunteers, With Contrast (N=8) | Patients With CKD III, With Contrast (N=66)
Chest pain (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Exacerbation of heart failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
2nd degree heart block (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Volunteers, no Contrast (N=8) | Volunteers With CKD III, no Contrast (N=8) | Healthy Volunteers, With Contrast (N=8) | Patients With CKD III, With Contrast (N=66)
Vomited (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vasovagal (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Chest pain (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bleeding from radial catheter site (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ischaemic ECG changes post-Angio (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Short self-terminating run of VT (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes